CLINICAL TRIAL: NCT06191744
Title: A Phase 3, Multicenter, Randomized, Open-Label Trial to Evaluate the Safety and Efficacy of Epcoritamab + Rituximab and Lenalidomide (R2) Compared to Chemoimmunotherapy in Previously Untreated Follicular Lymphoma (EPCORE™FL-2)
Brief Title: Study of Subcutaneous Epcoritamab in Combination With Intravenous Rituximab and Oral Lenalidomide (R2) to Assess Adverse Events and Change in Disease Activity in Adult Participants With Previously Untreated Follicular Lymphoma
Acronym: EPCORE™FL-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M22-003; 2023-506906-38-00 (Other: EU CT)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Follicular Lymphoma (FL)
Keywords: Follicular Lymphoma (FL); Non-Hodgkin's lymphoma (NHL); Lymphoma; Cancer; Epcoritamab; Rituximab; Lenalidomide; Chemoimmunotherapy (CIT); Obinutuzumab; Cyclophosphamide; Doxorubicin Hydrochloride; Vincristine Sulfate; Prednisone; Bendamustine (Benda); R-CHOP; G-CHOP; R-Benda; G-Benda; EPCORE™FL-2
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms | interventions — Prednisone; Rituximab; Lenalidomide; Doxorubicin; Vincristine; Cyclophosphamide; obinutuzumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Arm A1: Epcoritamab + Lenalidomide and Rituximab (R2) (Experimental): Participants will receive epcoritamab in combination with R2 (ER2), followed by epcoritamab during the 120 week treatment duration.
  Interventions: Drug: Epcoritamab; Drug: Rituximab; Drug: Lenalidomide
- Arm A2: Epcoritamab + Lenalidomide and Rituximab (R2) (Experimental): Participants will receive epcoritamab in combination with R2 (ER2), during the 24 week treatment duration.
  Interventions: Drug: Epcoritamab; Drug: Rituximab; Drug: Lenalidomide
- Arm B: Chemoimmunotherapy (CIT) Option A (Experimental): Participants will receive CIT Option A (obinutuzumab (G) and cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP) [G-CHOP]/ rituximab (R)-CHOP during the 120 week treatment duration.
  Interventions: Drug: Prednisone; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Obinutuzumab
- Arm B: Chemoimmunotherapy (CIT) Option B (Experimental): Participants will receive CIT Option B (G and bendamustine (Benda) [G-Benda]/R-Benda during the 120 week treatment duration.
  Interventions: Drug: Prednisone; Drug: Rituximab; Drug: Obinutuzumab; Drug: Bendamustine
- Arm C: Lenalidomide and Rituximab (R2) (Experimental): Participants will receive lenalidomide and rituximab (R2) during the 120 week treatment duration.
  Interventions: Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous (SC) Injection
  Other Names: ABBV-GMAB-3013; GEN3013; Epkinly
  Arms: Arm A1: Epcoritamab + Lenalidomide and Rituximab (R2); Arm A2: Epcoritamab + Lenalidomide and Rituximab (R2)
Drug: Prednisone — Oral Tablet
  Arms: Arm B: Chemoimmunotherapy (CIT) Option A; Arm B: Chemoimmunotherapy (CIT) Option B
Drug: Rituximab — Intravenous (IV) Infusion
Drug: Lenalidomide — Oral Capsule
  Arms: Arm A1: Epcoritamab + Lenalidomide and Rituximab (R2); Arm A2: Epcoritamab + Lenalidomide and Rituximab (R2); Arm C: Lenalidomide and Rituximab (R2)
Drug: Doxorubicin — IV Injection
  Arms: Arm B: Chemoimmunotherapy (CIT) Option A
Drug: Vincristine — IV Injection
  Arms: Arm B: Chemoimmunotherapy (CIT) Option A
Drug: Cyclophosphamide — IV Injection
  Arms: Arm B: Chemoimmunotherapy (CIT) Option A
Drug: Obinutuzumab — IV Infusion
  Arms: Arm B: Chemoimmunotherapy (CIT) Option A; Arm B: Chemoimmunotherapy (CIT) Option B
Drug: Bendamustine — IV Infusion
  Arms: Arm B: Chemoimmunotherapy (CIT) Option B

SUMMARY:
Follicular lymphoma (FL) is the second most common B-cell cancer and the most common type of cancer of lymphocytes. Unfortunately, this disease is incurable with conventional treatment and the disease recurs in almost all patients. This study will assess how safe and effective epcoritamab is in combination with lenalidomide and rituximab (R2) in treating adult participants with previously untreated FL. Adverse events and change in disease condition will be assessed.

Epcoritamab is an investigational drug being developed for the treatment of FL. Study doctors put the participants in 1 of 5 groups, called treatment arms. Each group receives a different treatment. Around 1095 adult participants with previously untreated FL will be enrolled in approximately 250 sites across the world.

Participants will receive R2 (intravenous [IV] infusion of rituximab (R) and oral capsules of lenalidomide) alone or in combination with subcutaneous injections of epcoritamab. Participants may also receive investigator's choice chemoimmunotherapy (CIT): IV infusion of obinutuzumab (G) and IV injections of cyclophosphamide, IV injections of doxorubicin, IV injections of vincristine, oral tablets of prednisone (CHOP) [G-CHOP]/ R-CHOP or G and IV infusion of bendamustine (Benda) [G-Benda]/R-Benda. The total treatment duration will be 120 weeks for all arms except A2, which is 24 weeks of treatment.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of follicular lymphoma (FL).
* Have CD20+, histologically confirmed classic FL (previously Grade 1 to 3a FL) at most recent representative tumor biopsy based on the local pathology report, according to the 5th edition of World Health Organization (WHO) Classification of Haematolymphoid Tumours.
* Are willing and able to comply with procedures required in the protocol.
* Must have stage, III, IV or II with bulky disease >= 7cm).
* Must be in need of systemic treatment per investigator, as evidenced by meeting at least one of the Groupe d'Etude des Lymphomes Folliculaire (GELF) criteria.
* Has one or more target lesions:

  * A positron emission tomography (PET)/computerized tomography (CT) scan demonstrating PET-positive lesion(s), and
  * >=1 measurable nodal lesion (long axis >1.5cm) or >=1 measurable extra-nodal lesion (long axis >1.0 cm) on CT scan or MRI
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Able to receive at least one of the standard of care chemoimmunotherapy (CIT) treatment regimens: [Arm B] at the discretion of the Investigator, and rituximab and lenalidomide (R2) [Arm C].
* Have laboratory values meeting the criteria in the protocol.

Exclusion Criteria:

* Had major surgery within 4 weeks prior to randomization.
* Have active cytomegalovirus (CMV) disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1095 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2037-11 (Estimated); Study Completion 2037-11 (Estimated)

PRIMARY OUTCOMES:
Arm A1 vs Arm B: Percentage of Participants who Achieve Complete Response rate at 30 months (CR30) | Up to 30 Months
  CR30 will be determined by positron emission tomography-computerized tomography (cat scan) [PET-CT] per Lugano 2014 criteria, as assessed by independent review committee (IRC).
Arm A1 vs Arm B: Number of Participants with Progression-free survival (PFS) | Up to 10 Years
  PFS is defined as the time from randomization until disease progression determined by Lugano 2014 criteria per IRC, or death, whichever occurs first.

SECONDARY OUTCOMES:
Arm A1 vs Arm B: Overall Survival (OS) | Up to 10 Years
  OS is defined as the time from the date of randomization to the date of death of any cause.
Arm A1 vs Arm B: Rate of Minimal Residual Disease (MRD) Negativity Rate | Up to 10 Years
  MRD negativity rate, defined as the absence of tumor specific molecules in whole blood and/or bone marrow in participants with follicular lymphoma (FL) MRD at baseline.
Arm A1 vs Arm B: Change from Baseline in Physical Functioning (PF) According to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer (EORTC QLQ-C30) | 21 Weeks
  The PF of EORTC QLQ-C30 is a 5-item questionnaire to assess the physical function of the participant, with a higher score indication worse functioning.
Arm A1 vs Arm A2: Percentage of Participants who Achieve CR30 | Up to 30 Months
  CR30 will be determined by PET-CT per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm C: Percentage of Participants who Achieve CR30 | Up to 30 Months
  CR30 will be determined by PET-CT per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm A2: Number of Participants with PFS | Up to 10 Years
  PFS is defined as the time from randomization until disease progression determined by Lugano 2014 criteria per IRC, or death, whichever occurs first.
Arm A1 vs Arm C: Number of Participants with PFS | Up to 10 Years
  PFS is defined as the time from randomization until disease progression determined by Lugano 2014 criteria per IRC, or death, whichever occurs first.
Arm A1 vs Arm A2: Rate of MRD Negativity | Up to 10 Years
  MRD negativity, defined as the absence of tumor specific molecules in whole blood and/or bone marrow in participants with FL MRD at baseline.
Arm A1 vs Arm C: Rate of MRD Negativity | Up to 10 Years
  MRD negativity, defined as the absence of tumor specific molecules in whole blood and/or bone marrow in participants with FL MRD at baseline.
Arm A1 vs Arm A2: Change from Baseline in PF According to EORTC QLQ-C30 | Up to 10 Years
  The PF of EORTC QLQ-C30 is a 5-item questionnaire to assess the physical function of the participant, with a higher score indication worse functioning.
Arm A1 vs Arm C: Change from Baseline in PF According to EORTC QLQ-C30 | Up to 10 Years
  The PF of EORTC QLQ-C30 is a 5-item questionnaire to assess the physical function of the participant, with a higher score indication worse functioning.
Arm A1 vs Arm A2: OS | Up to 10 Years
  OS is defined as the time from the date of randomization to the date of death of any cause.
Arm A1 vs Arm C: OS | Up to 10 Years
  OS is defined as the time from the date of randomization to the date of death of any cause.
Arm A1 vs Arm A2: Percentage of Participants who Achieve CR30 | Up to 30 Months
  CR30 will be determined by PET-CT per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm B: Percentage of Participants who Achieve CR30 | Up to 30 Months
  CR30 will be determined by PET-CT per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm C: Percentage of Participants who Achieve CR30 | Up to 30 Months
  CR30 will be determined by PET-CT per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm A2: Number of Participants with PFS | Up to 10 Years
  PFS is defined as the time from randomization until disease progression determined by Lugano 2014 criteria per investigator, or death, whichever occurs first.
Arm A1 vs Arm B: Number of Participants with PFS | Up to 10 Years
  PFS is defined as the time from randomization until disease progression determined by Lugano 2014 criteria per investigator, or death, whichever occurs first.
Arm A1 vs Arm C: Number of Participants with PFS | Up to 10 Years
  PFS is defined as the time from randomization until disease progression determined by Lugano 2014 criteria per investigator, or death, whichever occurs first.
Arm A1 vs Arm A2: Percentage of Participants with Change in CR Rate per IRC | Up to 10 Years
  CR will be determined by PET-CT per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm A2: Percentage of Participants with Change in CR Rate per Investigator | Up to 10 Years
  CR will be determined by PET-CT per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm B: Percentage of Participants with Change in CR Rate per IRC | Up to 10 Years
  CR will be determined by PET-CT per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm B: Percentage of Participants with Change in CR Rate per Investigator | Up to 10 Years
  CR will be determined by PET-CT per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm C: Percentage of Participants with Change in CR Rate per IRC | Up to 10 Years
  CR will be determined by PET-CT per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm C: Percentage of Participants with Change in CR Rate per Investigator | Up to 10 Years
  CR will be determined by PET-CT per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm A2: Number of Participants with Best Overall Response (BOR) per per Investigator | Up to 10 Years
  BOR is defined as the percentage of participants who achieve CR or partial response (PR) determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Arm A1 vs Arm A2: Number of Participants with BOR per IRC | Up to 10 Years
  BOR is defined as the percentage of participants who achieve CR or PR determined by Lugano 2014 criteria as assessed by IRC, or death from any cause.
Arm A1 vs Arm B: Number of Participants with BOR per Investigator | Up to 10 Years
  BOR is defined as the percentage of participants who achieve CR or PR determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Arm A1 vs Arm B: Number of Participants with BOR per IRC | Up to 10 Years
  BOR is defined as the percentage of participants who achieve CR or PR determined by Lugano 2014 criteria as assessed by IRC, or death from any cause.
Arm A1 vs Arm C: Number of Participants with BOR per Investigator | Up to 10 Years
  BOR is defined as the percentage of participants who achieve CR or PR determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Arm A1 vs Arm C: Number of Participants with BOR per IRC | Up to 10 Years
  BOR is defined as the percentage of participants who achieve CR or PR determined by Lugano 2014 criteria as assessed by IRC, or death from any cause.
Arm A1 vs Arm A2: Number of Participants with Event-free Survival (EFS) per IRC | Up to 10 Years
  EFS is defined as the time from randomization until adverse event determined by Lugano 2014 criteria per IRC, or death, whichever occurs first.
Arm A1 vs Arm A2: Number of Participants with EFS per Investigator | Up to 10 Years
  EFS is defined as the time from randomization until adverse event determined by Lugano 2014 criteria per investigator, or death, whichever occurs first.
Arm A1 vs Arm B: Number of Participants with EFS per IRC | Up to 10 Years
  EFS is defined as the time from randomization until adverse event determined by Lugano 2014 criteria per IRC, or death, whichever occurs first.
Arm A1 vs Arm B: Number of Participants with EFS per Investigator | Up to 10 Years
  EFS is defined as the time from randomization until adverse event determined by Lugano 2014 criteria per investigator, or death, whichever occurs first.
Arm A1 vs Arm C: Number of Participants with EFS per IRC | Up to 10 Years
  EFS is defined as the time from randomization until adverse event determined by Lugano 2014 criteria per IRC, or death, whichever occurs first.
Arm A1 vs Arm C: Number of Participants with EFS per Investigator | Up to 10 Years
  EFS is defined as the time from randomization until adverse event determined by Lugano 2014 criteria per investigator, or death, whichever occurs first.
Arm A1 vs Arm A2: Duration of Response (DOR) per IRC | Up to 10 Years
  DOR is defined as the time from PR or CR to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm A2: DOR per Investigator | Up to 10 Years
  DOR is defined as the time from PR or CR to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm B: DOR per IRC | Up to 10 Years
  DOR is defined as the time from PR or CR to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm B: DOR per Investigator | Up to 10 Years
  DOR is defined as the time from PR or CR to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm C: DOR per IRC | Up to 10 Years
  DOR is defined as the time from PR or CR to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm C: DOR per Investigator | Up to 10 Years
  DOR is defined as the time from PR or CR to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm A2: Duration of Complete Response (DOCR) per IRC | Up to 10 Years
  DOCR is defined as the time from CR to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm A2: DOCR per Investigator | Up to 10 Years
  DOCR is defined as the time from CR to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm B: DOCR per IRC | Up to 10 Years
  DOCR is defined as the time from CR to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm B: DOCR per Investigator | Up to 10 Years
  DOCR is defined as the time from CR to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm C: DOCR per IRC | Up to 10 Years
  DOCR is defined as the time from CR to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm C: DOCR per Investigator | Up to 10 Years
  DOCR is defined as the time from CR to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm A2: Time to Next Anti-lymphoma Therapy (TTNT) per Investigator | Up to 10 Years
  TTNT is defined as the time from randomization to first documented administration of subsequent anti-lymphoma therapy.
Arm A1 vs Arm A2: TTNT per IRC | Up to 10 Years
  TTNT is defined as the time from randomization to first documented administration of subsequent anti-lymphoma therapy.
Arm A1 vs Arm A2: TTNT per Investigator | Up to 10 Years
  TTNT is defined as the time from randomization to first documented administration of subsequent anti-lymphoma therapy.
Arm A1 vs Arm B: TTNT per IRC | Up to 10 Years
  TTNT is defined as the time from randomization to first documented administration of subsequent anti-lymphoma therapy.
Arm A1 vs Arm B: TTNT per Investigator | Up to 10 Years
  TTNT is defined as the time from randomization to first documented administration of subsequent anti-lymphoma therapy.
Arm A1 vs Arm C: TTNT per IRC | Up to 10 Years
  TTNT is defined as the time from randomization to first documented administration of subsequent anti-lymphoma therapy.
Arm A1 vs Arm C: TTNT per Investigator | Up to 10 Years
  TTNT is defined as the time from randomization to first documented administration of subsequent anti-lymphoma therapy.
Arm A1 vs Arm A2: Time to Progression per IRC | Up to 10 Years
  Time to progression defined as the time from randomization to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm A2: Time to Progression per Investigator | Up to 10 Years
  Time to progression defined as the time from randomization to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm B: Time to Progression per IRC | Up to 10 Years
  Time to progression defined as the time from randomization to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm B: Time to Progression per Investigator | Up to 10 Years
  Time to progression defined as the time from randomization to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm C: Time to Progression per IRC | Up to 10 Years
  Time to progression defined as the time from randomization to disease progression per Lugano 2014 criteria, as assessed by IRC.
Arm A1 vs Arm C: Time to Progression per Investigator | Up to 10 Years
  Time to progression defined as the time from randomization to disease progression per Lugano 2014 criteria, as assessed by investigator.
Arm A1 vs Arm A2: Number of Participants with Progression-free Survival After Subsequent Anti-Lymphoma Therapy (PFS2) | Up to 10 Years
  PFS2 is defined as the time after subsequent anti-lymphoma therapy to the earliest occurrence of disease progression determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Arm A1 vs Arm B: Number of Participants with PFS2 | Up to 10 Years
  PFS2 is defined as the time after subsequent anti-lymphoma therapy to the earliest occurrence of disease progression determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Arm A1 vs Arm C: Number of Participants with PFS2 | Up to 10 Years
  PFS2 is defined as the time after subsequent anti-lymphoma therapy to the earliest occurrence of disease progression determined by Lugano 2014 criteria as assessed by investigator, or death from any cause.
Arm A1 vs Arm A2: Change in Tolerability as Measured by Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 10 Years
  The PRO-CTCAE is a patient-reported outcome measurement system developed to assess symptomatic toxicity in participants in cancer clinical trials. PRO-CTCAE items evaluate common symptoms from study treatment on their frequency, severity, interference, amount, presence/absence.
Arm A1 vs Arm B: Change in Tolerability as Measured by PRO-CTCAE | Up to 10 Years
  The PRO-CTCAE is a patient-reported outcome measurement system developed to assess symptomatic toxicity in participants in cancer clinical trials. PRO-CTCAE items evaluate common symptoms from study treatment on their frequency, severity, interference, amount, presence/absence.
Arm A1 vs Arm C: Change in Tolerability as Measured by PRO-CTCAE | Up to 10 Years
  The PRO-CTCAE is a patient-reported outcome measurement system developed to assess symptomatic toxicity in participants in cancer clinical trials. PRO-CTCAE items evaluate common symptoms from study treatment on their frequency, severity, interference, amount, presence/absence.
Arm A1 vs Arm A2: Change in Tolerability as Measured by The Functional Assessment of Cancer Therapy - General (FACT-G) Item GP5 | Up to 10 Years
  The functional assessment of cancer therapy singly item - GP5 (FACT-GP5) is a single question asking if participant is bothered by side effects of treatment.
Arm A1 vs Arm B: Change in Tolerability as Measured by FACT-G Item GP5 | Up to 10 Years
  The FACT-GP5 is a single question asking if participant is bothered by side effects of treatment.
Arm A1 vs Arm C: Change in Tolerability as Measured by FACT-GG Item GP5 | Up to 10 Years
  The FACT-GP5 is a single question asking if participant is bothered by side effects of treatment.
Arm A1 vs Arm A2: Change in Symptoms as Measured by The Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) | Up to 10 Years
  The objective of the FACT-Lym patient reported outcome (PRO) is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm B: Change in Symptoms as Measured by FACT-Lym | Up to 10 Years
  The objective of the FACT-Lym patient reported outcome (PRO) is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm C: Change in Symptoms as Measured by FACT-Lym | Up to 10 Years
  The objective of the FACT-Lym patient reported outcome (PRO) is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm A2: Change in Quality of Life (QoL) as Measured by FACT-Lym | Up to 10 Years
  The objective of the FACT-Lym PRO is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm B: Change in QoL as Measured by FACT-Lym | Up to 10 Years
  The objective of the FACT-Lym PRO is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm C: Change in QoL as Measured by FACT-Lym | Up to 10 Years
  The objective of the FACT-Lym PRO is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm A2: Time-to-first PRO deterioration (TTD) in well-being using the lymphoma subscale (LymS) of FACT-Lym | Up to 10 Years
  The objective of the FACT-Lym PRO is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm B: TTD in well-being using LymS of FACT-Lym | Up to 10 Years
  The objective of the FACT-Lym PRO is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm C: TTD in well-being using LymS of FACT-Lym | Up to 10 Years
  The objective of the FACT-Lym PRO is to assess health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Likert-type scale.
Arm A1 vs Arm A2: Change in QoL as Measured by 5-Level European Quality of Life (EuroQol)-5-dimension [EQ-5D-5L] | Up to 10 Years
  The EQ-5D-5L is a standardized, non-disease specific instrument used to measure health-related quality of life. The EQ-5D-5L assesses general health on 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The scores for the 5 dimensions are used to compute a single utility index score ranging from 0 to 1 representing the general health status of the individual, with higher scores indicating better health state.
Arm A1 vs Arm B: Change in QoL as Measured by EQ-5D-5L | Up to 10 Years
  The EQ-5D-5L is a standardized, non-disease specific instrument used to measure health-related quality of life. The EQ-5D-5L assesses general health on 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The scores for the 5 dimensions are used to compute a single utility index score ranging from 0 to 1 representing the general health status of the individual, with higher scores indicating better health state.
Arm A1 vs Arm C: Change in QoL as Measured by EQ-5D-5L | Up to 10 Years
  The EQ-5D-5L is a standardized, non-disease specific instrument used to measure health-related quality of life. The EQ-5D-5L assesses general health on 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The scores for the 5 dimensions are used to compute a single utility index score ranging from 0 to 1 representing the general health status of the individual, with higher scores indicating better health state.
Arm A1 vs Arm A2: TTD in PF using the QLQ-C30 Physical Functioning Scale | Up to 10 Years
  The PF of EORTC QLQ-C30 is a 5-item questionnaire to assess the physical function of the participant, with a higher score indication worse functioning.
Arm A1 vs Arm B: TTD in PF using the QLQ-C30 Physical Functioning Scale | Up to 10 Years
  The PF of EORTC QLQ-C30 is a 5-item questionnaire to assess the physical function of the participant, with a higher score indication worse functioning.
Arm A1 vs Arm C: TTD in PF using the QLQ-C30 Physical Functioning Scale | Up to 10 Years
  The PF of EORTC QLQ-C30 is a 5-item questionnaire to assess the physical function of the participant, with a higher score indication worse functioning.
Arm A1 vs Arm A2: Change from baseline in the remaining items and domains of the EORTC QLQ-C30 | Up to 10 Years
  The EORTC QLQ-C30: A 30 items questionnaire to assess the quality of life of cancer patients on physical, emotional, cognitive, and social functions and symptoms. with a higher score indication worse quality of life.
Arm A1 vs Arm B: Change from baseline in the remaining items and domains of the EORTC QLQ-C30 | Up to 10 Years
  The EORTC QLQ-C30: A 30 items questionnaire to assess the quality of life of cancer patients on physical, emotional, cognitive, and social functions and symptoms. with a higher score indication worse quality of life.
Arm A1 vs Arm C: Change from baseline in the remaining items and domains of the EORTC QLQ-C30 | Up to 10 Years
  The EORTC QLQ-C30: A 30 items questionnaire to assess the quality of life of cancer patients on physical, emotional, cognitive, and social functions and symptoms. with a higher score indication worse quality of life.
Arm A1 vs Arm A2: Change in Patient Global Impression of Change (PGIC) for General Lymphoma Symptoms | Up to 10 Years
  The self-report measure PGIC reflects a participant's belief about the efficacy of treatment. The PGIC is a 7-point scale depicting a participant's rating of overall improvement since start of treatment. Participants rate their change as very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Arm A1 vs Arm C: Change in PGIC for General Lymphoma Symptoms | Up to 10 Years
  The self-report measure PGIC reflects a participant's belief about the efficacy of treatment. The PGIC is a 7-point scale depicting a participant's rating of overall improvement since start of treatment. Participants rate their change as very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Arm A1 vs Arm A2: Change in Patient Global Impression of Severity (PGIS) for General Lymphoma Symptoms | Up to 10 Years
  The self-report measure PGIS reflects a participant's belief about their lymphoma symptoms over the past 7 days. The PGIS is a 5-point scale depicting a participant's rating of overall severity.
Arm A1 vs Arm B: Change in PGIS for General Lymphoma Symptoms | Up to 10 Years
  The self-report measure PGIS reflects a participant's belief about their lymphoma symptoms over the past 7 days. The PGIS is a 5-point scale depicting a participant's rating of overall severity.
Arm A1 vs Arm C: Change in PGIS for General Lymphoma Symptoms | Up to 10 Years
  The self-report measure PGIS reflects a participant's belief about their lymphoma symptoms over the past 7 days. The PGIS is a 5-point scale depicting a participant's rating of overall severity.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (264):
- United States (57):
  - Scripps Mercy Hospital /ID# 265393, San Diego, California
  - Sansum Clinic Research /ID# 261596, Santa Barbara, California
  - Rocky Mountain Cancer Centers - Boulder /ID# 261203, Boulder, Colorado
  - Christiana Care Health Service /ID# 261207, Newark, Delaware
  - Cancer Specialists of North Florida - Jacksonville - AC Skinner Parkway /ID# 262445, Jacksonville, Florida
  - Advent Health /ID# 261578, Orlando, Florida
  - Orlando Health Cancer Institute /ID# 260983, Orlando, Florida
  - Moffitt Cancer Center /ID# 259487, Tampa, Florida
  - Beacon Cancer Care /ID# 260670, Coeur d'Alene, Idaho
  - Northwestern University- Robert H. Lurie Comprehensive Cancer Center /ID# 259814, Chicago, Illinois
  - Cancer Care Specialists Of Central Illinois /ID# 272464, Decatur, Illinois
  - Loyola University /ID# 259462, Maywood, Illinois
  - Illinois Cancer Care, PC /ID# 261526, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology- South Office /ID# 259583, Fort Wayne, Indiana
  - University of Iowa Health Care /ID# 262132, Des Moines, Iowa
  - University of Louisville Hospital /ID# 260544, Louisville, Kentucky
  - Norton Cancer Institute - St. Matthews /ID# 261076, Louisville, Kentucky
  - New England Cancer Specialists - Westbrook /ID# 260672, Westbrook, Maine
  - University of Maryland, Baltimore /ID# 259538, Baltimore, Maryland
  - Center for Cancer and Blood Disorders-American Oncology Partners of Maryland /ID# 259476, Bethesda, Maryland
  - St. Luke's Hospital - Chesterfield /ID# 260489, Chesterfield, Missouri
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana /ID# 260006, Billings, Montana
  - Nebraska Cancer Specialists (NCS) - Regional Cancer Center - St Francis Location /ID# 262506, Grand Island, Nebraska
  - NHO - Nebraska Hematology-Oncology /ID# 269692, Lincoln, Nebraska
  - Nebraska Cancer Specialists - Omaha - Wright Street /ID# 262505, Omaha, Nebraska
  - University of Nebraska Medical Center /ID# 261996, Omaha, Nebraska
  - University of New Mexico /ID# 261083, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital /ID# 262451, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center /ID# 262447, Rio Rancho, New Mexico
  - New York Oncology Hematology - Albany Cancer Center /ID# 261814, Albany, New York
  - NYU Langone Hospital - Long Island /ID# 265531, Mineola, New York
  - NYU Langone Medical Center /ID# 264518, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 259595, New York, New York
  - New York Oncology Hematology /ID# 270208, Troy, New York
  - Clinical Research Alliance, Inc. /ID# 261078, Westbury, New York
  - Novant Health Presbyterian Medical Center /ID# 259740, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center /ID# 259741, Winston-Salem, North Carolina
  - Oncology Hematology Care, Inc - Blue Ash /ID# 261204, Cincinnati, Ohio
  - Taylor Cancer Research Center /ID# 260488, Maumee, Ohio
  - Oncology Associates of Oregon, P.C. /ID# 261816, Eugene, Oregon
  - MUSC Hollings Cancer Center /ID# 259604, Charleston, South Carolina
  - Prisma Health /ID# 259602, Greenville, South Carolina
  - Sarah Cannon Research Institute - Tristar Centennial Medical Center /ID# 274985, Nashville, Tennessee
  - Texas Oncology - Austin Midtown /ID# 261208, Austin, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 261206, Dallas, Texas
  - MD Anderson Cancer Center /ID# 260984, Houston, Texas
  - Oncology Consultants /ID# 268390, Houston, Texas
  - Joe Arrington Cancer Research /ID# 260382, Lubbock, Texas
  - Intermountain Healthcare LDS Hospital /ID# 259759, Salt Lake City, Utah
  - Virginia Cancer Specialists - Fairfax /ID# 261205, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia /ID# 261592, Roanoke, Virginia
  - Swedish Cancer Institute - Edmonds /ID# 266356, Edmonds, Washington
  - Swedish Cancer Institute - Issaquah /ID# 266358, Issaquah, Washington
  - Vista Oncology - East Olympia /ID# 261360, Olympia, Washington
  - Virginia Mason Hospital & Medical Center /ID# 260549, Seattle, Washington
  - Swedish Cancer Institute /ID# 260370, Seattle, Washington
  - Northwest Medical Specialties - Tacoma /ID# 262133, Tacoma, Washington
- Australia (10):
  - Royal Prince Alfred Hospital /ID# 259320, Camperdown, New South Wales
  - Liverpool Hospital /ID# 259321, Liverpool, New South Wales
  - Peter MacCallum Cancer Center /ID# 260431, Melbourne, New South Wales
  - Westmead Hospital /ID# 261465, Westmead, New South Wales
  - Townsville University Hospital /ID# 259323, Douglas, Queensland
  - Royal Brisbane and Women's Hospital /ID# 259326, Herston, Queensland
  - Princess Alexandra Hospital /ID# 259329, Woolloongabba, Queensland
  - Peninsula Private Hospital /ID# 259325, Frankston, Victoria
  - Fiona Stanley Hospital /ID# 259324, Murdoch, Western Australia
  - Royal Perth Hospital /ID# 259319, Perth, Western Australia
- Belgium (7):
  - Algemeen Ziekenhuis klina /ID# 260324, Brasschaat, Antwerpen
  - Uza /Id# 260319, Edegem, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 260311, Brussels, Brussels Capital
  - Groupe Sante CHC - Clinique du MontLegia /ID# 260325, Liège, Liege
  - UZ Gent /ID# 260312, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 260304, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 260313, Roeselare, West-Vlaanderen
- Brazil (9):
  - Oncocentro de Minas Gerais /ID# 260973, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaertner /ID# 260871, Curitiba, Puerto Rico
  - Hospital Amaral Carvalho - Fundacao Doutor Amaral Carvalho /ID# 260828, Jaú, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 260843, Ribeirão Preto, São Paulo
  - Fundacao Antonio Prudente - AC Camargo Cancer Center /ID# 260827, São Paulo, São Paulo
  - Grupo Oncoclínicas Botafogo /ID# 260870, Rio de Janeiro
  - Real e Benemérita Associação Portuguesa de Beneficência /ID# 260826, São Paulo
  - Instituto D'Or de Pesquisa e Ensino - Regional Sao Paulo /ID# 260829, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 260822, São Paulo
- Bulgaria (4):
  - UMHAT Dr Georgi Stranski EAD /ID# 260763, Pleven
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 260685, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 259277, Sofia
  - SHAT Hematologic Diseases /ID# 260457, Sofia
- Canada (5):
  - Victoria Hospital /ID# 260770, London, Ontario
  - The Ottawa Hospital - General Campus /ID# 264470, Ottawa, Ontario
  - CSSS Alphonse-Desjardins, CHAU de Levis /ID# 260527, Lévis, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM) /ID# 260617, Montreal, Quebec
  - Disc_Royal Victoria Hospital / McGill University Health Centre /ID# 261075, Montreal, Quebec
- China (28):
  - Peking University First Hospital /ID# 259816, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 259806, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University /ID# 260014, Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center /ID# 260478, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital /ID# 260446, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University /ID# 260558, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 260795, Guangzhou, Guangdong
  - Shenzhen People's Hospital /ID# 260137, Shenzhen, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University /ID# 260537, Nanning, Guangxi
  - People's Hospital of Henan Province /ID# 259619, Zhengzhou, Henan
  - Henan Cancer Hospital /ID# 259618, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 259743, Wuhan, Hubei
  - Hubei Cancer Hospital /ID# 260506, Wuhan, Hubei
  - Hunan Cancer Hospital /ID# 260439, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University /ID# 260507, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 260556, Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital /ID# 260559, Nanchang, Jiangxi
  - First Affiliated Hospital of China Medical University /ID# 260217, Shenyang, Liaoning
  - Shandong Cancer Hospital /ID# 260808, Jinan, Shandong
  - Fudan University Cancer Hospital /ID# 260564, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 260015, Chengdu, Sichuan
  - Tianjin Cancer Hospital /ID# 259807, Tianjin, Tianjin Municipality
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 259616, Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital of Xinjiang Medical University /ID# 260644, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital /ID# 260645, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 259744, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital /ID# 259742, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 260566, Wenzhou, Zhejiang
- Croatia (7):
  - Clinical Hospital Dubrava /ID# 260452, Zagreb, City of Zagreb
  - Klinicka bolnica Merkur /ID# 260393, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 260456, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 260364, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka /ID# 260455, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 260454, Split, Split-Dalmatia County
  - Zadar General Hospital /ID# 260837, Zadar
- Czechia (3):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 260571, Brno, Brno-mesto
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 260560, Hradec Králové, Hradec Kralove
  - Fakultni nemocnice Kralovske Vinohrady /ID# 260572, Prague
- Denmark (5):
  - Rigshospitalet /ID# 260779, Copenhagen Ø, Capital Region
  - Regionshospitalet Godstrup /ID# 260778, Herning, Central Jutland
  - Roskilde Sygehus /ID# 260780, Roskilde, Region Sjælland
  - Odense University Hospital /ID# 260777, Odense, Region Syddanmark
  - Vejle Sygehus /ID# 260781, Vejle, Region Syddanmark
- France (10):
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 260875, Caen, Calvados
  - CHU Brest - Hôpital de la Cavale Blanche /ID# 260601, Brest, Finistere
  - Hopital Prive du Confluent /ID# 260596, Nantes, Loire-Atlantique
  - Centre Hospitalier D'Avignon /ID# 260511, Avignon, Provence-Alpes-Côte d'Azur Region
  - HCL - Hopital Lyon Sud /ID# 260508, Pierre-Bénite, Rhone
  - Centre Hospitalier du Mans /ID# 260510, Le Mans, Sarthe
  - CH Libourne - Hopital Robert Boulin /ID# 261478, Libourne
  - Hôpital Saint-Louis /ID# 260509, Paris
  - Clinique Sainte-Anne /ID# 261528, Strasbourg
  - Hopital Prive d'Antony /ID# 260598, Antony, Île-de-France Region
- Germany (6):
  - Staedtisches Klinikum Karlsruhe /ID# 260348, Karlsruhe, Baden-Wurttemberg
  - Universitaetsklinikum Frankfurt /ID# 260388, Frankfurt am Main, Hesse
  - Klinikum Kassel /ID# 260432, Kassel, Hesse
  - St.-Antonius-Hospital /ID# 260520, Eschweiler, North Rhine-Westphalia
  - Klinikum Ludwigshafen /ID# 260688, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Otto-von-Guericke-Universitaet /ID# 260425, Magdeburg, Saxony-Anhalt
- Greece (5):
  - Olympion General Clinic /ID# 262395, Pátrai, Achaia
  - General Hospital of Athens Laiko /ID# 259708, Athens, Attica
  - University General Hospital Attikon /ID# 260855, Athens, Attica
  - General University Hospital of Alexandroupolis /ID# 260858, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 259709, Athens
- Hungary (5):
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz /ID# 260051, Győr, Győr-Moson-Sopron
  - Tolna Varmegyei Balassa Janos Korhaz /ID# 260048, Szekszárd, Tolna County
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 260050, Szombathely, Vas County
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 260049, Budapest
  - Orszagos Onkologiai Intezet /ID# 260052, Budapest
- Israel (7):
  - Meir Medical Center /ID# 259938, Kfar Saba, Central District
  - HaEmek Medical Center /ID# 259936, Afula, Haifa District
  - Hadassah /ID# 259935, Jerusalem, Jerusalem
  - Soroka University Medical Center /ID# 259937, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 259934, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 259933, Tel Aviv, Tel Aviv
  - Rabin Medical Center. /ID# 268328, Petah Tikva
- Italy (7):
  - IRCCS Istituto Clinico Humanitas /ID# 260887, Rozzano, Lombardy
  - Istituto di Candiolo Fondazione del Piemonte per l'Oncologia IRCCS /ID# 260889, Candiolo, Torino
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 260886, Bologna
  - AOU Policlinico G. Rodolico - San Marco /ID# 260890, Catania
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 260888, Palermo
  - AUSL di Reggio Emilia - Arcispedale Santa Maria Nuova /ID# 260744, Reggio Emilia
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 260891, Roma
- Japan (21):
  - Fujita Health University Hospital /ID# 264679, Toyoake, Aichi-ken
  - Matsuyama Red Cross Hospital /ID# 266426, Matsuyama, Ehime
  - University of Fukui Hospital /ID# 265680, Yoshida-gun, Fukui
  - National Hospital Organization Kyushu Cancer Center /ID# 265960, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 267861, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 264994, Fukushima, Fukushima
  - Chugoku Central Hospital /ID# 266520, Fukuyama, Hiroshima
  - Sapporo Medical University Hospital /ID# 265031, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital /ID# 266379, Kobe, Hyōgo
  - Hitachi General Hospital /ID# 265676, Hitachi-shi, Ibaraki
  - Kitasato University Hospital /ID# 264675, Sagamihara-shi, Kanagawa
  - Kanagawa Cancer Center /ID# 265497, Yokohama, Kanagawa
  - Okayama University Hospital /ID# 267135, Okayama, Okayama-ken
  - Kansai Medical University Hospital /ID# 266019, Hirakata-shi, Osaka
  - Kindai University Hospital /ID# 265038, Sakai-shi, Osaka
  - Tokyo Metropolitan Komagome Hospital /ID# 267692, Bunkyo Ku, Tokyo
  - The University of Tokyo Hospital /ID# 266422, Bunkyo-ku, Tokyo
  - Yamaguchi University Hospital /ID# 265619, Ube, Yamaguchi
  - University of Yamanashi Hospital /ID# 264677, Chuo-shi, Yamanashi
  - Aomori Prefectural Central Hospital /ID# 265692, Aomori
  - Chiba Cancer Center /ID# 267316, Chiba
- Netherlands (9):
  - Bravis Ziekenhuis /ID# 259055, Bergen op Zoom, North Brabant
  - Elisabeth Tweesteden Ziekenhuis /ID# 261239, Tilburg, North Brabant
  - Olvg /Id# 259543, Amsterdam, North Holland
  - Leids Universitair Medisch Centrum /ID# 259049, Leiden, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis /ID# 259052, Rotterdam, South Holland
  - HagaZiekenhuis /ID# 261220, The Hague, South Holland
  - St. Antonius Ziekenhuis /ID# 259053, Nieuwegein, Utrecht
  - Rijnstate /ID# 261219, Arnhem
  - Universitair Medisch Centrum Groningen /ID# 259051, Groningen
- New Zealand (2):
  - Auckland City Hospital /ID# 259330, Grafton, Auckland
  - North Shore Hospital /ID# 260824, Takapuna, Auckland
- Poland (5):
  - Aidport sp z o.o. /ID# 267717, Poznan, Greater Poland Voivodeship
  - Pratia MCM Krakow /ID# 260075, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. M. Sklodowskiej /ID# 260861, Warsaw, Masovian Voivodeship
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopern /ID# 260633, Lodz, Łódź Voivodeship
  - Swietokrzyskie Centrum Onkologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej /ID# 260170, Kielce, Świętokrzyskie Voivodeship
- Portugal (4):
  - Fundacao Champalimaud /ID# 259652, Lisbon, Lisbon District
  - Unidade Local de Saude de Gaia/Espinho, EPE /ID# 259655, Vila Nova de Gaia, Porto District
  - Unidade Local de Saude de Santa Maria, EPE /ID# 259650, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE /ID# 259649, Porto
- Puerto Rico (2):
  - Pan American Center for Oncology Trials, LLC /ID# 260265, Rio Piedras
  - Auxilio Mutuo Cancer Center /ID# 260262, San Juan
- Romania (4):
  - Fundeni Clinical Institute /ID# 260296, Bucharest, București
  - Institutul Oncologic Prof Dr. Ion Chiricuta Cluj Napoca /ID# 259704, Cluj-Napoca, Cluj
  - Institutul Regional de Oncologie /ID# 259697, Iași, Iaşi
  - Spitalul Clinic Coltea /ID# 259699, Bucharest
- Serbia (5):
  - Clinical Hospital Center Zvezdara /ID# 260900, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 259271, Belgrade, Beograd
  - University Clinical Center Kragujevac /ID# 259274, Kragujevac, Sumadijski Okrug
  - Institute for Oncology of Vojvodina /ID# 260223, Kamenitz, Vojvodina
  - University Clinical Center Vojvodina /ID# 259272, Novi Sad
- Slovakia (2):
  - Narodny onkologicky ustav /ID# 260638, Bratislava, Bratislava Region
  - Univerzitna nemocnica Martin /ID# 260631, Martin, Žilina Region
- South Africa (3):
  - Wits Clinical Research /ID# 260958, Johannesburg, Gauteng
  - Alberts Cellular Therapy /ID# 260514, Pretoria, Gauteng
  - Haemalife Inc. /ID# 260513, Kuils River, Western Cape
- South Korea (4):
  - Seoul National University Bundang Hospital /ID# 260009, Seongnam-si, Gyeonggido
  - Seoul National University Hospital /ID# 260007, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 260010, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 260008, Seoul, Seoul Teugbyeolsi
- Spain (11):
  - Instituto Catalan de Oncologia (ICO) Badalona /ID# 260495, Badalona, Barcelona
  - Institut Català d'Oncologia (ICO) - L'Hospitalet /ID# 261439, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla /ID# 260497, Santander, Cantabria
  - Clinica Universidad de Navarra - Pamplona /ID# 260496, Pamplona, Navarre
  - Hospital Universitario Vall de Hebron /ID# 260490, Barcelona
  - Hospital Clinic de Barcelona /ID# 260492, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 260498, Barcelona
  - Hospital San Pedro de Alcantara /ID# 260502, Cáceres
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 261512, Madrid
  - MD Anderson Madrid /ID# 260500, Madrid
  - Hospital Universitario de Salamanca /ID# 260491, Salamanca
- Sweden (2):
  - Sodra Alvsborgs sjukhus /ID# 261168, Borås, Västra Götaland County
  - Sahlgrenska Universitetssjukhuset /ID# 266600, Gothenburg, Västra Götaland County
- Taiwan (4):
  - National Taiwan University Hospital /ID# 260341, Taipei City, Taipei
  - China Medical University Hospital /ID# 260357, Taichung
  - Taichung Veterans General Hospital /ID# 260361, Taichung
  - National Cheng Kung University Hospital /ID# 260363, Tainan
- Turkey (Türkiye) (5):
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 259804, Istanbul
  - Ege Universitesi Tip Fakultesi /ID# 259803, Izmir
  - Kocaeli University Med Faculty /ID# 259717, Kocaeli
  - Ondokuz Mayis Universitesi /ID# 259713, Samsun
  - Istanbul Florence Nightingale Hospital /ID# 271291, Şişli
- United Kingdom (6):
  - Derriford Hospital and the Royal Eye Infirmary /ID# 262671, Plymouth, Devon
  - Hammersmith Hospital /ID# 261124, London, England
  - Queen Alexandra Hospital /ID# 269708, Portsmouth, Hampshire
  - Leeds Teaching Hospitals NHS Trust /ID# 260466, Leeds, West Yorkshire
  - The Christie Hospital /ID# 260463, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 260792, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-003